CLINICAL TRIAL: NCT02713412
Title: Cardiovascular Function and Postprandial Hypotension (PPH): Effect of an Oral Glucose Load on Cardiac Contractility, Cardiac Output, Diastolic Function and Endothelial Function - Relationship to Gastric Emptying
Brief Title: Effects of Water and Glucose Drinks on Cardiovascular Function in Subjects With and Without Postprandial Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Responsible Party: Principal Investigator, Karen Jones, Professor, Royal Adelaide Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HREC/12/TQEHLMH/106
Record Dates: First submitted 2016-03-06; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Autonomic Nervous System Diseases; Baroreflex Failure; Blood Pressure; Hypotension
MeSH Terms: conditions — Autonomic Nervous System Diseases; Hypotension | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose (Experimental): 75g glucose and 150mg C13-acetate in 300ml water
  Interventions: Other: Glucose
- Control (Placebo Comparator): 300ml water
  Interventions: Other: Water

INTERVENTIONS:
Other: Glucose — 75g glucose and 150 mg of 13C-acetate made up to 300 ml with water
  Arms: Glucose
Other: Water — 300ml water
  Arms: Control

SUMMARY:
To determine whether the changes in blood pressure (BP) which occur following meals in normal people and patients who have substantial falls in BP after a meal postprandial hypotension (PPH)) are associated with changes in cardiac function. Eligible subjects who have been previously diagnosed with PPH will report to the Queen Elizabeth Hospital, on two occasions, following an overnight fast. Subjects will be cannulated and have a BP cuff placed around their upper arm. Following this, subjects will ingest either a drink containing 75 grams of glucose and 150mg of a C13 Acetate (which is metabolised and excreted in the breath, enabling noninvasive measurements of gastric emptying), made up to 300mL water, or on the other study day, 300mL water alone. The order of the study days will be randomised. Following the drink, for 3 hours, measurements will be taken at regular intervals of BP, heart rate, breath samples (on the study day with the Acetate only), blood samples (for measurement of blood glucose and gut hormones) and transthoracic echocardiography (TTE) (for assessment of end systolic and diastolic cardiac volume, cardiac output, cardiac contractility and diastolic function). After the 3 hours of measurements, the cannula will be removed and subjects will be offered lunch prior to leaving the department. Following lunch, on one study day, subjects will have their autonomic nerve function tested noninvasively, using an ECG.

DETAILED DESCRIPTION:
Subjects who meet the inclusion criteria will be required to attend the Queen Elizabeth Hospital, on two separate occasions, at 08:30h following an overnight fast (solids for 14 hours and liquids for 12 hours) and abstaining from smoking for 12 hours prior to the study day. The order of the study days will be randomized using the online Random Integer Set Generator program (RANDOM.ORG).

On each of the study days, subjects will be seated and have an intravenous cannula inserted into an antecubital vein in the arm for blood sampling and an automated blood pressure (BP) cuff (DINAMAP ProCare 100, GE Medical Systems, Milwaukee, WI, USA) placed around the opposite arm for measurements of BP (systolic and diastolic) and heart rate (HR).

After a 15-minute rest period, subjects will consume a drink consisting of either 75g glucose and 150 mg of 13C-acetate made up to 300 ml with water, or 300 ml water, within 3 minutes (t = -3 - 0 minutes).

BP and HR will be measured at 3 minute intervals during the 30-minute rest period prior to the drink (i.e. t = -30 - 0 minutes) and at 3 minute intervals from t = 0 - 180 minutes.

Blood samples (~ 18ml) will be taken prior (t = -3 minutes) to the drink and then at t = 30, 60, 90, 120 and 180 minutes for the subsequent measurement of blood glucose, serum insulin and incretin hormones. Samples will be stored at -70°C until analysed. Blood glucose will be determined immediately using a portable glucometer (Medisense Companion 2 meter, Medisense Inc, Waltham, USA).

Following the 75g drink consisting of 75g glucose and 150 mg of 13C-acetate made up to 300 ml with water, at t = -3 minutes, and every 5 minutes between t = 0 - 60, followed by every 15 minutes between t = 60 - 180, breath samples will be collected in sealed tubes for subsequent analysis of 13CO2 for measurement of gastric emptying.

At t = -30 minutes and then at t = 30, 60, 90, 120 and 180 minutes, subjects will also undergo Transthoracic Echocardiogram (TTE) for assessment of (i) end-systolic and diastolic volumes (ii) cardiac output (iii) cardiac contractility, as assessed by measuring

1. left ventricular dP/dt and
2. overall wall motion by Doppler tissue imaging (DTI) of basal mitochondrial segments (iv) diastolic function, as assessed by measuring

a) mitral inflow velocities b) DTI of mitral annulus c) left atrial size and d) pulmonary vein flow patterns Prior to each measurement, subjects will be allowed to rest for 15 minutes, remaining still in a supine position.

At t = 180 the cannulae will be removed and subjects will be offered a light lunch before leaving the department. The total amount of blood collected during the two visits is ~180 ml.

On one of the study days after completion of these measurements autonomic nerve function will be assessed using standardised cardiovascular reflex tests. Parasympathetic function will be calculated by the variation (R - R interval) of the HR during deep breathing and the immediate HR response to standing ("30:15" ratio). Sympathetic function will be assessed by the fall in systolic BP in response to standing.

ELIGIBILITY:
Inclusion Criteria:

* Control subjects: subjects from this group will be healthy, with normal BMI. PPH subjects: Patients who have been diagnosed with PPH (defined as a fall in systolic blood pressure (BP) of > 20mmHg within 2 hours of a meal).

Exclusion Criteria:

* No history of severe respiratory, cardiovascular, hepatic and/or renal disease, diabetes, are not taking any medication with effects on blood pressure or gastrointestinal function, have not donated blood for the past 12 weeks or been involved in any research projects for the past 3 months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure over time. | time= 0 - 120 min
  time= 0 min is defined as the consumption of either the experimental or control drink, i.e. outcome will be assessed for 2 hours.

SECONDARY OUTCOMES:
Change from baseline cardiac output as assessed by echocardiography, over time. | time= 0 - 120 min
  time= 0 min is defined as the consumption of either the experimental or control drink, i.e. outcome will be assessed for 2 hours.
Change from baseline stroke volume as assessed by echocardiography, over time. | time= 0 - 120 min
  time= 0 min is defined as the consumption of either the experimental or control drink, i.e. outcome will be assessed for 2 hours.
Change from baseline ejection fraction as assessed by echocardiography, over time. | time= 0 - 120 min
  time= 0 min is defined as the consumption of either the experimental or control drink, i.e. outcome will be assessed for 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Jones, PhD, Principal Investigator — karen.jones@adelaide.edu.au

IPD SHARING:
Plan to Share IPD: Yes
Anonymous study data (minus all demographic data which compromises confidentiality) will be made available in a publicly accessible depository after publication.

REFERENCES:
- [Background] Gentilcore D, Nair NS, Vanis L, Rayner CK, Meyer JH, Hausken T, Horowitz M, Jones KL. Comparative effects of oral and intraduodenal glucose on blood pressure, heart rate, and splanchnic blood flow in healthy older subjects. Am J Physiol Regul Integr Comp Physiol. 2009 Sep;297(3):R716-22. doi: 10.1152/ajpregu.00215.2009. Epub 2009 Jun 24. PMID 19553500
- [Background] Jones KL, Tonkin A, Horowitz M, Wishart JM, Carney BI, Guha S, Green L. Rate of gastric emptying is a determinant of postprandial hypotension in non-insulin-dependent diabetes mellitus. Clin Sci (Lond). 1998 Jan;94(1):65-70. doi: 10.1042/cs0940065. PMID 9505868
- [Background] O'Donovan D, Feinle C, Tonkin A, Horowitz M, Jones KL. Postprandial hypotension in response to duodenal glucose delivery in healthy older subjects. J Physiol. 2002 Apr 15;540(Pt 2):673-9. doi: 10.1113/jphysiol.2001.013442. PMID 11956353
- [Background] Trahair LG, Vanis L, Gentilcore D, Lange K, Rayner CK, Horowitz M, Jones KL. Effects of variations in duodenal glucose load on blood pressure, heart rate, superior mesenteric artery blood flow and plasma noradrenaline in healthy young and older subjects. Clin Sci (Lond). 2012 Mar;122(6):271-9. doi: 10.1042/CS20110270. PMID 21942924
- [Background] Vanis L, Gentilcore D, Hausken T, Pilichiewicz AN, Lange K, Rayner CK, Feinle-Bisset C, Meyer JH, Horowitz M, Jones KL. Effects of gastric distension on blood pressure and superior mesenteric artery blood flow responses to intraduodenal glucose in healthy older subjects. Am J Physiol Regul Integr Comp Physiol. 2010 Sep;299(3):R960-7. doi: 10.1152/ajpregu.00235.2010. Epub 2010 Jun 16. PMID 20554933
- [Background] Braden B, Adams S, Duan LP, Orth KH, Maul FD, Lembcke B, Hor G, Caspary WF. The [13C]acetate breath test accurately reflects gastric emptying of liquids in both liquid and semisolid test meals. Gastroenterology. 1995 Apr;108(4):1048-55. doi: 10.1016/0016-5085(95)90202-3. PMID 7698571
- [Background] Chew CG, Bartholomeusz FD, Bellon M, Chatterton BE. Simultaneous 13C/14C dual isotope breath test measurement of gastric emptying of solid and liquid in normal subjects and patients: comparison with scintigraphy. Nucl Med Rev Cent East Eur. 2003;6(1):29-33. PMID 14600930
- [Background] Mossi S, Meyer-Wyss B, Beglinger C, Schwizer W, Fried M, Ajami A, Brignoli R. Gastric emptying of liquid meals measured noninvasively in humans with [13C]acetate breath test. Dig Dis Sci. 1994 Dec;39(12 Suppl):107S-109S. doi: 10.1007/BF02300386. PMID 7995201
- [Background] Piha SJ. Cardiovascular autonomic reflex tests: normal responses and age-related reference values. Clin Physiol. 1991 May;11(3):277-90. doi: 10.1111/j.1475-097x.1991.tb00459.x. PMID 1893685